CLINICAL TRIAL: NCT03910387
Title: Weight Loss in Patients With Advanced Stage Pancreatic Cancer: Role of Serotonin and Effects of Telotristat Ethyl
Brief Title: Telotristat Ethyl to Promote Weight Stability in Patients With Advanced Stage Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lexicon Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Olumide Gbolahan, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00105292; NCI-2018-01977 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4441-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Unresectable Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Recurrent Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; telotristat ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) (Experimental): Patients receive gemcitabine/nab-paclitaxel combination chemotherapy on days 1, 8 and 15, and telotristat ethyl PO QD, BID, or TID on days 1 and 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Telotristat Ethyl
- Group 2 (gemcitabine/nab-paclitaxel) (Active Comparator): Patients receive gemcitabine/nab-paclitaxel chemotherapy (at the discretion of the investigator) on days 1, 8 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Given gemcitabine/nab-paclitaxel combination therapy
  Other Names: Gemzar; dFdCyd; Difluorodeoxycytidine
Drug: Nab-paclitaxel — Given gemcitabine/nab-paclitaxel combination therapy
  Other Names: ABI-007; Abraxane; Nanoparticle Albumin-bound Paclitaxel
Drug: Telotristat Ethyl — Given PO
  Other Names: Xermelo
  Arms: Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl)

SUMMARY:
This phase II trial studies how well telotristat ethyl works in promoting weight stability in patients with pancreatic adenocarcinoma that has come back and spread to other places in the body. Telotristat ethyl may decrease bowel movements which may make patients gain weight. Stabilizing weight may help patients tolerate chemotherapy better and improve longevity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate weight stability after 3 months of telotristat ethyl treatment in patients who have significant weight loss (documented to be more than or equal to 10%) prior to the start of treatment. (Group 1).

II. Evaluate the change in serum and 24-hours (hr) urine 5-hydroxyindoleacetic acid (5-HIAA) in patients with locally advanced unresectable, recurrent or metastatic pancreatic adenocarcinoma (PDAC) receiving chemotherapy. (Group 2).

SECONDARY OBJECTIVES:

I. Evaluate the impact of weight stabilization/gain on patients in Group 1 on performance status, quality of life (QOL), mid arm circumference (MAC) and muscle mass on cross sectional imaging.

II. Evaluate correlations between changes in serotonin/ 5HIAA levels on radiologic response, weight stability, mid arm circumference (MAC), and muscle mass on cross sectional imaging.

III. Evaluate the relation of baseline serum and 24-hr urine 5-HIAA on weight loss in patients with advanced PDAC.

IV. Safety and tolerability of telotristat ethyl with gemcitabine/nab-paclitaxel combination chemotherapy.

V. Evaluate response rate (RR) assessed per Response Evaluation Criteria in Solid Tumors (RECIST), progression free survival and overall survival in patients receiving telotristat ethyl (Group 1).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1: Patients receive gemcitabine/nab-paclitaxel combination chemotherapy on days 1, 8 and 15, and telotristat ethyl orally (PO) once daily (QD), twice daily (BID), or thrice daily (TID) on days 1 and 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP 2: Patients receive chemotherapy (at the discretion of the investigator) on days 1, 8 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* GROUP 1 (Telotristat ethyl treatment group): Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* GROUP 1 (Telotristat ethyl treatment group): Weight loss of 10% or more.
* GROUP 1 (Telotristat ethyl treatment group): Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 within 14 days prior to registration.
* GROUP 1 (Telotristat ethyl treatment group): Histologic or cytological diagnosis of recurrent or metastatic pancreas adenocarcinoma (PDAC) who present for first line chemotherapy treatment for metastatic disease.
* GROUP 1 (Telotristat ethyl treatment group): Advanced stage pancreas cancer (recurrent/metastatic).
* GROUP 1 (Telotristat ethyl treatment group): Measurable disease determined using guidelines of Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Baseline tumor assessment should be performed using high resolution computed tomography (CT) scans or magnetic resonance imaging (MRI).
* GROUP 1 (Telotristat ethyl treatment group): Prior systemic therapy (adjuvant or neoadjuvant setting are acceptable) if disease progressed or recurred within at least 3 months after treatment.
* GROUP 1 (Telotristat ethyl treatment group): Estimated life expectancy of > 12 weeks, as assessed by the site investigator.
* GROUP 1 (Telotristat ethyl treatment group): If sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods) due to unknown risk of teratogenicity.
* GROUP 1 (Telotristat ethyl treatment group): Hemoglobin ≥ 8 g/dL (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Absolute Neutrophil Count (ANC) ≥ 1,500/mm³ (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Platelet Count (PLT) ≥ 100,000/mm³ (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Creatinine ≤ 1.5 mg/dL (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Albumin ≥ 2 g/dL (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Bilirubin ≤ 1.5 mg/dL (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN) or < 5 x ULN in the setting of liver metastases (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Alanine aminotransferase (ALT) ≤ 3 x ULN or < 5 x ULN in the setting of liver metastases (obtained within 7 days prior to registration).
* GROUP 1 (Telotristat ethyl treatment group): Prior radiation is allowed if happened more than 2 weeks of enrollment.
* GROUP 2 (Non-Telotristat ethyl group): Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* GROUP 2 (Non-Telotristat ethyl group): Stable weight or loss of < 10% by history.
* GROUP 2 (Non-Telotristat ethyl group): ECOG Performance Status of 0-2 within 14 days prior to registration.
* GROUP 2 (Non-Telotristat ethyl group): Histologic or cytological diagnosis of locally advanced unresectable, recurrent/metastatic PDAC who present for first line chemotherapy treatment for metastatic disease.
* GROUP 2 (Non-Telotristat ethyl group): Advanced stage PDAC (locally advanced unresectable/recurrent/metastatic).
* GROUP 2 (Non-Telotristat ethyl group): Prior systemic therapy (adjuvant or neoadjuvant setting are acceptable) if disease progressed or recurred within at least 3 months after treatment.
* GROUP 2 (Non-Telotristat ethyl group): Estimated life expectancy of > 12 weeks, as assessed by the site investigator.
* GROUP 2 (Non-Telotristat ethyl group): Prior radiation is allowed if happened more than 2 weeks of enrollment.

Exclusion Criteria:

* GROUP 1 (Telotristat ethyl treatment group): Subjects with histology other than adenocarcinoma. Examples include: neuroendocrine tumors, acinar cell cancer, sarcoma or lymphoma of the pancreas.
* GROUP 1 (Telotristat ethyl treatment group): Ongoing or active infection.
* GROUP 1 (Telotristat ethyl treatment group): Symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia. Symptomatic heart failure (New York Heart Association [NYHA] Class II-IV).
* GROUP 1 (Telotristat ethyl treatment group): Acute or sub-acute intestinal obstruction.
* GROUP 1 (Telotristat ethyl treatment group): Ascites.
* GROUP 1 (Telotristat ethyl treatment group): Documented and/or symptomatic or known brain or leptomeningeal metastases.
* GROUP 1 (Telotristat ethyl treatment group): Severely immune-compromised (other than being on steroids) including known human immunodeficiency virus (HIV) infection.
* GROUP 1 (Telotristat ethyl treatment group): Concurrent active malignancy, other than adequately treated non-melanoma skin cancer, other noninvasive carcinoma, or in situ neoplasm. A subject with previous history of malignancy is eligible if he/she has been disease-free for > 3 years.
* GROUP 1 (Telotristat ethyl treatment group): Breast-feeding or pregnant. Serum pregnancy test for women of child-bearing potential must be performed within 7 days prior to first dose of study treatment.
* GROUP 1 (Telotristat ethyl treatment group): Prior autologous or allogeneic organ or tissue transplantation.
* GROUP 1 (Telotristat ethyl treatment group): Known allergy to any of the treatment components.
* GROUP 1 (Telotristat ethyl treatment group): Have any condition that does not permit compliance with the study schedule including psychological, geographical, or medical.
* GROUP 1 (Telotristat ethyl treatment group): Not able to swallow. Inability to take oral medications.
* GROUP 1 (Telotristat ethyl treatment group): Patients with chronic constipation.
* GROUP 2 (Non-Telotristat ethyl group): Subjects with histology other than adenocarcinoma. Examples include: neuroendocrine tumors, acinar cell cancer, sarcoma or lymphoma of the pancreas.
* GROUP 2 (Non-Telotristat ethyl group): Ongoing or active infection.
* GROUP 2 (Non-Telotristat ethyl group): Symptomatic congestive heart failure, unstable angina or arrhythmia. Symptomatic heart failure (NYHA Class II-IV).
* GROUP 2 (Non-Telotristat ethyl group): Acute or sub-acute intestinal obstruction.
* GROUP 2 (Non-Telotristat ethyl group): Severely immune-compromised (other than being on steroids) including known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gehan Botrus, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Started | 14 | 9
Completed | 14 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Gemcitabine/Nab-paclitaxel and Telotristat Ethyl) | Group 2 (Gemcitabine/Nab-paclitaxel) | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Weight Stability
Description: Weight stability will be documented as percent weight change at 3 months compared to baseline.
Time Frame: Baseline up to 3 months after study start
Measure: Mean (Standard Deviation); unit: Percent weight change
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 14 | 8
Percent weight change | -1.98 (6.87) | -5.58 (5.89)

2. Secondary Outcome: Change in 24-hr Urine 5-hydroxyindoleacetic Acid (5-HIAA) Levels
Description: The change will be summarized as mean and standard deviation.
Time Frame: Baseline up to 4 months after study start
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 10 | 5
Milligrams
  Screening | 3 (261.67) | 4 (46.25)
  Cycle 1 Day 1 (Treatment day 0) | 8 (232.38) | 3 (44.87)
  Cycle 2 Day 1 (Treatment day 28) | 8 (58.63) | 2 (144.00)
  Cycle 3 Day 1 (Treatment day 56) | 7 (119.10) | 1 (273.00)
  Cycle 4 Day 1 (Treatment day 84) | 9 (91.56) | 1 (10.00)

3. Secondary Outcome: Mid Arm Circumference (MAC) Measured in cm
Description: Mid arm circumference (MAC) will be reviewed on cross sectional imaging and will be assessed with imaging guided measurements of the psoas and rectus abdominis muscle.
Time Frame: Up to 2 years after study start
Population: This OC was not collected at the following timepoints, and a protocol amendment did not occur.
  Cycle 7 Day 1, Group 2 Cycle 8 Day 1, Group 2 Cycle 10 Day 1, Group 1 Cycle 11 Day 1, Group 1 Cycle 12 Day 1, Group 1 Cycle 13 Day 1, Group 1 Cycle 14 Day 1, Group 1 Cycle 15 Day 1, Group 1 & 2 Cycle 17 Day 1, Group 1 &2 Cycle 18 Day 1 Group 2 Cycle 19 Day 1, Group 2 Cycle 22 Day 1, Group 2 Cycle 23 Day 1, Group 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 14 | 5
cm
  Screening: number analyzed (Participants) | 11 | 4
  Screening | 24.35 (9.43) | 34.88 (6.17)
  Cycle 1 Day 1: number analyzed (Participants) | 11 | 4
  Cycle 1 Day 1 | 24.39 (8.69) | 35.88 (5.86)
  Cycle 2 Day 1: number analyzed (Participants) | 9 | 3
  Cycle 2 Day 1 | 23.98 (7.28) | 35.5 (5.89)
  Cycle 3 Day 1: number analyzed (Participants) | 9 | 1
  Cycle 3 Day 1 | 25.71 (6.12) | 27 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 4 Day 1: number analyzed (Participants) | 9 | 2
  Cycle 4 Day 1 | 25.71 (6.52) | 29 (7.07)
  Cycle 5 Day 1: number analyzed (Participants) | 3 | 2
  Cycle 5 Day 1 | 24.81 (3.52) | 31.5 (0.71)
  Cycle 6 Day 1: number analyzed (Participants) | 4 | 1
  Cycle 6 Day 1 | 26.67 (6.24) | 31 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 7 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 7 Day 1 | 27.81 (4.52) |
  Cycle 8 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 8 Day 1 | 21.81 (8.59) |
  Cycle 9 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 9 Day 1 | 25.4 (NA) — Only 1 participant analyzed. SD is NA. | 29 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 10 Day 1 |  | 30 (0)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 11 Day 1 |  | 30 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 12 Day 1 |  | 30 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 13 Day 1 |  | 26 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 14 Day 1 |  | 24 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 16 Day 1 | 29.21 (NA) — Only 1 participant analyzed. SD is NA. |
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 18 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 18 Day 1 | 23 (NA) — Only 1 participant analyzed. SD is NA. |
  Cycle 19 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 19 Day 1 | 25 (NA) — Only 1 participant analyzed. SD is NA. |
  Cycle 20 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 20 Day 1 | 23 (NA) — Only 1 participant analyzed. SD is NA. |
  Cycle 21 Day 1: number analyzed (Participants) | 1 | 1
  Cycle 21 Day 1 | 26 (NA) — Only 1 participant analyzed. SD is NA. | 24.5 (NA) — Only 1 participant analyzed. SD is NA.
  Cycle 22 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 22 Day 1 | 25 (NA) — Only 1 participant analyzed. SD is NA. |
  Cycle 23 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 23 Day 1 | 28.5 (NA) — Only 1 participant analyzed. SD is NA. |

4. Secondary Outcome: Quality of Life (QOL)
Description: Quality of life (QOL) will be assessed by the Obesity Related Quality of Life (OWL-QOL)-17 questionnaire.
  *Please note OC Measure was not collected.
Time Frame: Up to 2 years after study start
Reporting Status: Not Posted

5. Secondary Outcome: Blood Serotonin Levels
Description: Blood serotonin levels will be compared in the 2 groups.
Time Frame: Up to 2 years after study start
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 14 | 8
ng/mL
  Screening | 170.92 [121.02 to 220.82] | 294.67 [213.97 to 375.37]
  Cycle 1 Day 1 (Treatment day 0 | 152.75 [106.58 to 198.92] | 201.33 [191.89 to 228.77]
  Cycle 2 Day 1 (Treatment day 28) | 96.09 [56.73 to 135.45] | 217 [183.48 to 250.52]
  Cycle 3 Day 1 (Treatment day 56) | 97.67 [54.05 to 141.29] | 112.67 [34.29 to 191.05]
  Cycle 4 Day 1 (Treatment day 84) | 85.33 [53.51 to 117.15] | 265 [0 to 1531.81]

6. Secondary Outcome: Response Rate (RR)
Description: Response rate (RR) will be assessed per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, in patients receiving telotristat ethyl (Group 1).
Time Frame: Up to 2 years after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 12 | 6
Participants | 11 | 6

7. Secondary Outcome: Median Overall Survival (MOS)
Description: Median overall survival (MOS) will be measured using the Kaplan-Meier method.
Time Frame: Up to 2 years after study start
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 14 | 8
Days | 10.7 [5.4 to 16.9] | 12.2 [6.1 to 21.4]

8. Secondary Outcome: Duration of Response
Description: Duration of response will be estimated from time of documentation of response to time of progression and will be evaluated by computed tomography/magnetic resonance imaging scans of the organ(s) with the target lesion(s) based on RECIST criteria.
Time Frame: Up to 2 years after study start
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
Number analyzed (Participants) | 9 | 6
Days | 94 [9 to 172] | 97 [60 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) | Group 2 (gemcitabine/nab-paclitaxel)
All-Cause Mortality (participants affected / at risk) | 9/14 | 6/8
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/8
Other Adverse Events (participants affected / at risk) | 13/14 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) (N=14) | Group 2 (gemcitabine/nab-paclitaxel) (N=8)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (gemcitabine/nab-paclitaxel and telotristat ethyl) (N=14) | Group 2 (gemcitabine/nab-paclitaxel) (N=8)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (24) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (17) | 1 (1)
General disorders and administration site conditions (General disorders) | 9 (20) | 1 (11)
Infections and infestations (Infections and infestations) | 0 (0) | 1 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Investigations (Investigations) | 4 (52) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 (23) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 4 (9) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 2 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Vascular disorders (Vascular disorders) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03910387/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03910387/ICF_001.pdf